CLINICAL TRIAL: NCT00020787
Title: An Open Label, Sequential Multi-Center Multi Dose Study Of G17T Immunogen In Combination With Cisplatin (CDDP) And 5-Fluorouracil (5-FU) In Subjects With Metastatic Or Locally Recurrent Gastric Or Gastroesophageal Cancer Previously Untreated With Chemotherapy For Advanced Disease (Stage IV)
Brief Title: Vaccine Therapy Plus Chemotherapy in Treating Patients With Metastatic or Locally Recurrent Stomach Cancer or Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Randolph Hecht, MD, UCLA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068713; UCLA-0006040; APHTON-BB-IND-8737; NCI-G01-1959; UCLA-GC4C
Record Dates: First submitted 2001-07-11; First posted 2004-01-08 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — gastrin immunogen; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See intervention description.
  Interventions: Biological: G17DT Immunogen; Drug: cisplatin; Drug: fluorouracil

INTERVENTIONS:
Biological: G17DT Immunogen — Dose: 500 micrograms in 0.2mL Route: Deep intramuscular Schedule: Days 8, 36, and 64; an additional dose at week 2, cycle 7 will be administered
Drug: cisplatin — dose: 100 mg/m2 Route: i.v. infusion in 500 mL in 0.9% NaCl administered up to 3 hours Schedule: day 1, and then every 4 weeks.
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II)
Drug: fluorouracil — Dose: 1000mg/m2/day Route: 24-hour continuous infusion in 0.9% NaCl over 5 days Schedule: Day 1 to Day 5 (5-day infusion) and then every 4 weeks
  Other Names: 5-FU

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy and chemotherapy in treating patients who have metastatic or locally recurrent stomach cancer or esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine a safe and immunogenic combination of G17DT with cisplatin and fluorouracil in patients with chemotherapy-naive metastatic or locally recurrent gastric or gastroesophageal cancer. II. Determine the safety profile and tolerability of this regimen in these patients. III. Determine the tumor response rate, disease stabilization, best overall response, time to progression, time to treatment failure, and overall survival in patients treated with this regimen. IV. Determine the correlation of immunological response with clinical efficacy and benefit in patients treated with this regimen. V. Determine the pharmacokinetics and pharmacodynamics of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are assigned to one of four treatment regimens. Regimen A: Patients receive high-dose G17DT intramuscularly (IM) on days 7, 35, and 63. Patients also receive cisplatin IV over 1-3 hours on day 1 followed by fluorouracil IV continuously over days 1-5 every 4 weeks in the absence of disease progression or unacceptable toxicity. If inadequate immune response is seen on Regimen A, subsequent patients are treated on Regimen B. If unacceptable toxicity is seen on Regimen A, subsequent patients are treated on Regimen C. If inadequate immune response and unacceptable toxicity are seen on Regimen A, or if unacceptable toxicity is seen on Regimen B or inadequate immune response is seen on Regimen C, then subsequent patients are treated on Regimen D. Regimen B: Patients receive high-dose G17DT IM on days 1, 28, and 56. Patients also receive cisplatin IV over 1-3 hours on day 35 followed by fluorouracil IV continuously over days 35-39 every four weeks in the absence of disease progression or unacceptable toxicity. Regimen C: Patients receive low-dose G17DT IM on days 7, 35, and 63 with chemotherapy as in regimen A. Regimen D: Patients receive low-dose G17DT IM on days 1, 28, and 56 with chemotherapy as in regimen B. Quality of life is assessed at baseline, on day 7, every 2 weeks for 10 weeks, and then every 4 weeks thereafter.

PROJECTED ACCRUAL: A total of 15-75 patients will be accrued for this study within 5-30 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Gastric adenocarcinoma, including adenocarcinoma of the esophagogastric junction, histologically proven.
* Measureable metastatic disease.
* Male or female subjects, age 18 years and older.
* Karnofsky performance status score equal to or greater than 70.
* Life expectancy of at least 3 months.
* Subjects must be chemotherapy naïve.
* At least 6 weeks from prior curative radiotherapy and 3 weeks from surgery.
* Adequate hematological and coagulation parameters: hemoglobin>9.5 g/dL; white blood cell count>3x10^9/L, platelets> 100x10^9/L; international normalized ratio of prothrombin time <1.2, and activated partial thromboplastin time no more than 5 seconds above normal limits.
* Adequate clinical chemistry parameters: creatinine<1.5mg/dL; total bilirubin<1.5mg/dL; and aspartate aminotransferase and alanine aminotransferase <2.5x upper normal levels.
* Able to comply with scheduled follow-up and with management of toxicity.
* Use contraceptive measures, if sexually active

Exclusion Criteria:

* Previous or current malignancies other than gastric adenocarcinoma, with the exception of adequately treated in situ carcinoma of the cervix, uteri, or nonmelanoma skin cancer
* Female subjects who are pregnant or nursing
* Female subjects with reproductive potential refusing a pregnancy test
* Any previous palliative chemotherapy, adjuvant or neoadjuvant chemotherapy, or investigational drug
* Any prior anticancer immunotherapy
* Immunodeficiency
* Bone marrow transplantation within 1 year
* Symptomatic peripheral neuropathy > Grade 2 NCI-CTC, Version 2.0 criteria
* Severe hearing disorder > Grade 2 NCI-CTC, Version 2.0 criteria
* Known dihydropyrimidine dehydrogenase deficiency
* Any other sever condition as defined by the following: unstable cardiac disease despite treatment; myocardial infarction within 6 months before study entry; history of significant neurologic or psychiatric disorders including dementia or seizures; active uncontrolled infection; active disseminated intravascular coagulation; or any other serious underlying medical conditions that could impair the ability of the subject to participate in the study
* Subjects who have previously demonstrated hypersensitivity to diphtheria toxoid
* Subjects who require chronic administration of corticosteroids
* Use in the past 30 days or concomitant use of immunosuppressants
* Use in the past 14 days or chronic concomitant use of proton pump inhibitors
* Subjects who have a history of hypercalcemia
* Subjects who cannot be regularly followed up for psychological, social, familial, or geographic reasons
* Subjects with expected noncompliance to toxicity management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2001-07; Primary Completion 2002-01 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
To determine whether a concomitant G17DT-chemotherapy regimen affects tumor response in subjects with gastric or gastroesophageal cancer. | 6 months to 1 year

SECONDARY OUTCOMES:
Time to disease progression, best overall response, and survival will be evaluated in the intent-to-treat population and the evaluable population. | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joel R. Hecht, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Ajani JA, Hecht JR, Ho L, Baker J, Oortgiesen M, Eduljee A, Michaeli D. An open-label, multinational, multicenter study of G17DT vaccination combined with cisplatin and 5-fluorouracil in patients with untreated, advanced gastric or gastroesophageal cancer: the GC4 study. Cancer. 2006 May 1;106(9):1908-16. doi: 10.1002/cncr.21814. PMID 16568451
- [Result] Hecht JR, Ajani JA, Michaeli D: A multicenter phase II study of cisplatin (CDDP) and 5-fluorouracil (5-FU) in combination with G17DT immunogen in patients with locally recurrent or metastatic adenocarcinoma of the stomach or gastroesophageal junction previously untreated for advanced disease. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1035, 258, 2003.